CLINICAL TRIAL: NCT02660190
Title: Photodynamic Diagnosis (PDD) in Flexible Cystoscopy - DaBlaCa-11
Brief Title: Photodynamic Diagnosis (PDD) in Flexible Cystoscopy
Acronym: DaBlaCa-11
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jørgen Bjerggaard Jensen (Other)
Collaborators: Regional Hospital West Jutland (Other); Herlev Hospital (Other)
Responsible Party: Sponsor-Investigator, Jørgen Bjerggaard Jensen, Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EudraCT no.: 2015-000
Record Dates: First submitted 2016-01-14; First posted 2016-01-21 (Estimated); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Bladder Cancer; Recurrence; PDD
MeSH Terms: conditions — Urinary Bladder Neoplasms; Recurrence | interventions — 5-aminolevulinic acid hexyl ester

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PDD (Experimental): PDD at flexible cystoscopy
  Interventions: Drug: hexaminoavolunate; Procedure: WL cystoscopy
- WL (Experimental): WL only at flexible cystoscopy
  Interventions: Procedure: WL cystoscopy

INTERVENTIONS:
Drug: hexaminoavolunate
  Other Names: hexvix
  Arms: PDD
Procedure: WL cystoscopy

SUMMARY:
Photodynamic diagnostic (PDD) is a technique where a photodynamic drug is installed preoperatively in the bladder. Mucosa cells with a higher metabolism than normal urothelial cells, e.g. cancer cells, absorbs this drug which is utilized during cystoscopy where blue light is absorbed by the drug, making the surgeon able to distinguish tumor cells from normal cells and thus being able to identify flat lesions and small papillomas missed in white light cystoscopy.

The use of PDD at this primary transurethral resection of bladder tumour (TURB) has been shown to be associated with a lower recurrence rate within the first year, probably mostly owing to a higher detection rate of small papillomas and dysplasia that therefore can be relevantly treated at an early stage.

Despite the use of PDD at the primary TURB, a high number of patients experience an early recurrence and patients with carcinoma in situ (CIS) treated with bacillus Calmette-Guerin (BCG) may have recurrence of their CIS or recurrence of papillomas despite the peroperative use of PDD.

Whereas the use of PDD is well established in the TURB setting, the use of PDD in the follow-up setting with flexible cystoscopy in the outpatient clinic is not investigated. Feasibility studies have been successful but the clinical relevance and benefits have not been investigated so far.

Thesis The thesis of the study is that the use of PDD in the outpatient clinic in patients with a high recurrence risk undergoing follow-up flexible cystoscopy will result in diagnosis of papillomas earlier than by the use of conventional flexible cystoscopy in white light. Thus, a higher number of tumours can be treated in the outpatient setting without the need for procedures in general anesthesia. Furthermore, the number of follow-up cystoscopies can be reduced if PDD is used at the first cystoscopy following TURB.

Aims To investigate whether the use of PDD when performing a flexible cystoscopy in the outpatient clinic can reduce the number of recurrences of large size papillomas that cannot be treated by simple fulguration without general anesthesia. Furthermore, to investigate whether the use of PDD in follow-up cystoscopy in patients with earlier complete response to BCG on CIS, can increase the detection rate of CIS recurrences.

DETAILED DESCRIPTION:
Background Bladder cancer is a very heterogeneous disease ranging from minimal pathology in small non-invasive Ta-tumors of low malignancy (Papillary Urothelial Neoplasm of Low Malignant Potential or low grade Ta tumours) easily fulgurated upon cystoscopy to deeply invasive metastasizing disease with fatal course despite aggressive treatment. Moreover, urothelial pathology ranges from flat lesions not visible in regular white light to massive bulky tumors.

In advanced tumor stages with deeply invasive T1-tumours or muscle invasive disease (T2) the highest risk is progression is tumour, nodes, metastases (TNM) stage and the largest challenge thus to prevent this with aggressive radical treatment. In the lowest tumor stages with non-invasive Ta-tumors and even superficially infiltrating non-muscle invasive tumors, the vast majority of patients do not progress regarding stage but more than half of the patients experience a recurrence of tumor at the same stage in the bladder. These recurrences are time consuming, expensive to treat because of the high number, and is affecting quality of life because they result in a need for frequent follow-up visits and recurrent procedures. Flat lesions recur frequently after intravesical treatment and is associated with a high risk of progression if left untreated.

Recurrent tumors are mostly treated by a transurethral resection of the bladder (TURB) in general anesthesia. However, if recognized at a very early stage, these tumors can be safely fulgurated in the outpatient clinic. Moreover, the recognition of flat lesions or even carcinoma in situ (CIS) at an earlier stage is presumed to be associated with a lower risk of progression to more advanced tumor stages.

Therefore, a reduction of the size and number of recurrences and early recognition of flat lesions is desired.

Early recurrences within the first year following the primary TURB are thought to arise in small areas of flat dysplasia, CIS, or small sub-visible papillomas not recognized at the primary procedure.

PDD is a technique where a photodynamic drug is installed preoperatively in the bladder. Mucosa cells with a higher metabolism than normal urothelial cells, e.g. cancer cells, absorbs this drug which is utilized during cystoscopy where blue light is absorbed by the drug, making the surgeon able to distinguish tumor cells from normal cells and thus being able to identify flat lesions and small papillomas missed in white light cystoscopy.

The use of PDD at this primary TURB has been shown to be associated with a lower recurrence rate within the first year, probably mostly owing to a higher detection rate of small papillomas and dysplasia that therefore can be relevantly treated at an early stage.

Despite the use of PDD at the primary TURB, a high number of patients experience an early recurrence and patients with carcinoma in situ (CIS) treated with bacillus Calmette-Guerin (BCG) may have recurrence of their CIS or recurrence of papillomas despite the peroperative use of PDD.

Whereas the use of PDD is well established in the TURB setting, the use of PDD in the follow-up setting with flexible cystoscopy in the outpatient clinic is not investigated. Feasibility studies have been successful but the clinical relevance and benefits have not been investigated so far.

Thesis The thesis of the study is that the use of PDD in the outpatient clinic in patients with a high recurrence risk undergoing follow-up flexible cystoscopy will result in diagnosis of papillomas earlier than by the use of conventional flexible cystoscopy in white light. Thus, a higher number of tumours can be treated in the outpatient setting without the need for procedures in general anesthesia. Furthermore, the number of follow-up cystoscopies can be reduced if PDD is used at the first cystoscopy following TURB.

Aims To investigate whether the use of PDD when performing a flexible cystoscopy in the outpatient clinic can reduce the number of recurrences of large size papillomas that cannot be treated by simple fulguration without general anesthesia.

Methods

The study is designed as a prospective, randomized study with randomization between conventional white light flexible cystoscopy or PDD flexible cystoscopy. The study includes the following category of patients that have the highest risk of tumor recurrence:

• All patients coming for first outpatient flexible cystoscopy 4 month after TURB without subsequent BCG instillations.

Patients will be informed of the study before the visit and if patient accept is given, randomization will be made at the time of cystoscopy. Patients in the PDD-arm will receive the intravesical instillation of Hexvix 1 hour prior of cystoscopy. Cystoscopy will be made with the Storz flexible PDD-cystoscope.

Patients will be handled and followed according to the national Danish bladder tumor guidelines. This includes follow-up cystoscopy 4 and 12 months following the primary TURB in patients with low grade Ta tumors and follow-up cystoscopy at four months interval the first 2 years following diagnosis in patients with high grade tumors or CIS. If tumor recurrence is diagnosed, size of the largest tumor is estimated based on the intervals: less than 5 mm, 5-10 mm, 11-20 mm, and more than 20 mm. All tumor recurrences and suspicious areas in the mucosa will be histologically verified either by resection or biopsy before fulguration.

Follow-up cystoscopies in the outpatient clinic are performed in white light (WL) in both arms.

Primary endpoint:

• Tumor recurrence found in outpatient flexible cystoscopies following but not including the cystoscopy 4 months after TURB where intervention is made. Patients are dichotomized regarding recurrence as primary endpoint in "any recurrence at any cystoscopy" versus "no recurrences" at cystoscopy 8 or 12 months of the primary TURB.

Secondary outcomes:

* Number of procedures in general anesthesia within 12 months of the TURB
* Tumor recurrence of more than 5 mm, 10 mm, and more than 20 mm within 12 months of the TURB
* Progression in stage within 12 months of the TURB
* Identification of flat lesions including CIS

Statistics Power calculation is made as one-sided testing at a 5% significance level with risk of type I error (alpha) of 0.05 and risk of type II error (beta) of 0.20. Given a recurrence rate of 35% within the first 12 month and presuming 15% of all patients have recurrence found at the 4 months cystoscopy leaves at minimum 20% for detection at 8 and 12 months cystoscopy. This recurrence rate s slightly underestimated because patients with recurrences after 4 months also have a high risk of recurrence at the following cystoscopies. Recurrence rate is estimated to be reduced by one third (absolute 7%) to 13 % at the 8 and 12 months cystoscopy by the use of PDD at 4 months cystoscopy. Thus, a number of 696 patients is needed when using equal sized groups of 348 in each of the randomization arms.

Ethics The study has been approved by the Regional Science Ethics Committee (Number 1-10-72-76-15) and the Danish Data Protection Agency (Number 1-16-02-111-15). The study will be reported on clinicaltrials.gov before initiation. The study has been submitted for approval at the Danish Health And Medicines Authority. The local good clinical practice (GCP)-units will be allocated to the trial.

Timeframe The study is planned to begin February 2016. Inclusion of patients all 696 patients is expected to be terminated within an 18 month period. Follow-up of the last patient included can be made 8 months following the inclusion giving an estimated time of study analysis in the end of 2018.

Set-up The study will be performed as a single surgeon, multi center study. Thus, one surgeon will be performing all cystoscopies at all three locations. Moreover the nurses involved in handling the cystoscopes and patients at each of the three locations will be limited to two at each location. This is to ensure the quality of the study and especially to reduce the risk of unintentional damage to the equipment including the cystoscopes.

The three study locations will be:

* The outpatient clinic in Herlev at Herlev Hospital
* The outpatient clinic in Holstebro at Hospital of West Denmark
* The outpatient clinic at Aarhus University Hospital Based on patient catchment area of the involved centers, it is expected to include 40% at Herlev Hospital (approximately 280 patients), 35% at Aarhus University Hospital (approximately 245 patients), and 25% at Hospital of West Denmark (approximately 175 patients). These are expected numbers subject to changes and will depend on inclusion rates at the involved centers.

Additional project regarding health economics, logistics and time used for flexible PDD Along with the major project, two additional projects will be performed. One is a research year student looking at health economics by using flexible PDD. In this, time spend for the additional examination and biopsy will be compared to the time saved in case of a reduced recurrence rate leading to fewer TURB's and cystoscopies. Moreover, the finances saved by reducing the number of TURB's and cystoscopies will be compared with the additional cost by using PDD. The other project is a nurse led study evaluating the feasibility and logistics by implementing flexible PDD in the outpatient clinic. These studies will be evaluating all three involved clinics to give a more valid insight than one-center studies.

ELIGIBILITY:
Inclusion Criteria:

* All patients coming for first outpatient flexible cystoscopy 4 month after TURB without subsequent BCG instillations

Exclusion Criteria:

* Muscle invasive bladder cancer (MIBC)
* BCG treatment within the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 696 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Tumor recurrence | 8 months
  Tumor recurrence up to 8 months following first cystoscopy after TURB

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Herlev Hospital, Herlev
  - Hospitalsenheden Vest, Holstebro

IPD SHARING:
Plan to Share IPD: No